CLINICAL TRIAL: NCT06484647
Title: Comparing T-stenting And Minimal Protrusion With External Minicrush for Treatment of Complex Coronary Bifurcation: Insights From TREX Registry
Brief Title: Comparing T-stenting And Minimal Protrusion With External Minicrush for Treatment of Complex Coronary Bifurcation
Status: Recruiting | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Medical Doctor, MD, San Luigi Gonzaga Hospital
Other Study IDs: 001-2024
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Chronic Coronary Syndrome; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention (PCI); Coronary Artery Disease (CAD); Coronary Bifurcation Lesion (CBL)
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T-stenting And Minimal Protrusion: Percutaneous coronary intervention is performing according to current coronary Revascularization guidelines (ACC/ESC).
  The vascular access is chosing according patients characteristics and operator preferences and require radial or femoral insertion of the sheath.
  Antiplatelets strategy is a discretion of the operator and is depending on clinical presentation of the patients and respect the current guidelines (i.e Clopidogrel 600 mg load dose following 75 mg/daily, Ticagrelor 180 mg load dose following 180 mg/daily, Prasugrel 60 mg load dose following 10 mg/daily).
  The procedural steps of the technique are described below:
  * MV stenting
  * Distal rewiring towards SB
  * Kissing Balloon for opening distal struts towards SB
  * SB stent implantation
  * Final Kissing Balloon
  Interventions: Procedure: Percutaneous Coronary Intervention
- External Minicrush: Percutaneous coronary intervention is performing according to current coronary Revascularization guidelines (ACC/ESC).
  The vascular access is chosing according patients characteristics and operator preferences and require radial or femoral insertion of the sheath.
  Antiplatelets strategy is a discretion of the operator and is depending on clinical presentation of the patients and respect the current guidelines (i.e Clopidogrel 600 mg load dose following 75 mg/daily, Ticagrelor 180 mg load dose following 180 mg/daily, Prasugrel 60 mg load dose following 10 mg/daily).
  The procedural steps of the technique are described below:
  * SB stent deployment with protrusion into MB
  * Crush the SB stent with a balloon inflating into MB (>0.5 mm of the SB stent)
  * MB stent deployment
  * Rewiring
    * POT
    * KBI
    * Final POT technique
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention is a procedure that require coronary stenosis dilatation with dilatation catheter balloon and generally stent implantation.
  The study involve coronary stenosis at bifurcation level that require complex coronary techniques such as External Minicrush or TAP technique.

SUMMARY:
Nowadays, no studies compare the T-stenting And Minimal Protrusion (TAP) and External Minicrush techniques in treating complex coronary bifurcation, so eventually, procedural, clinical and safety differences remain unknown.

DETAILED DESCRIPTION:
1. According to DEFINITION criteria, PCI of the complex coronary bifurcation with up-front two stent techniques is associated with lower target vessel revascularization (TVR) compared to Provisional Stenting
2. The Double-Kissing Crush stenting (DK-Crush) has been tested with the Culotte and the Classic Crush techniques in the unprotected left main disease (ULMD) and in no-ULMD setting, respectively, showing better clinical outcomes.
3. However, due to its technical complexity and simultaneous improvement of the Classic Crush technique evolving in the External Minicrush, it has meant that the latter has become the most used technique in the clinical practice in treating complex coronary bifurcation
4. The DK-Crush technique has never been tested with the External Minicrush, leaving the operators to choose one or the other according to their experience and preferences.
5. The T-stenting And Minimal Protrusion (TAP) is a two-stent technique described to treat coronary bifurcation after provisional treating. Compared to crush techniques, it does not require crushing of the side branch stent but only minimal protrusion of the side branch stent before main vessel stenting.
6. Nowadays, no studies compare theTAP and the External Minicrush in treating complex coronary bifurcation, so eventually, procedural, clinical and safety differences remain unknown.
7. The issue's importance is highlighted by higher rates of stent thrombosis (ST) and in-stent restenosis (ISR) of the two stent techniques compared to Provisional Stenting in treating coronary bifurcation8.
8. Consequently, investigating the efficacy and safety differences between the techniques could improve the treatment of complex coronary bifurcation to reduce post-PCI TLR.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Patients with an indication for PCI, including chronic coronary syndrome and acute coronary syndromes (STEMI, NSTEMI, unstable angina)
* Patients with at least one true coronary bifurcation according to the Medina classification 1.1.1, 0.1.1, 1.0.1, 0.0.1

Exclusion Criteria:

* Patients who do not want or cannot sign the informed consent for the procedure.
* Patients with severe peripheral vascular disease that limits vascular access to the point of making the procedure unsafe.
* Patients with a life expectancy of <1 year.
* Patients with planned major surgery require prolonged discontinuation of antiplatelet therapy.
* Pregnant women.
* Patients who cannot take antiplatelet therapy for any reason.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ACS or CCS patients with complex coronary bifurcation lesions with the indication of PCI.
Sampling Method: Non-Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 5-years
  a composite of cardiac death and target vessel-related myocardial infarction (TV-MI), including Q wave, non-Q wave myocardial infarction (MI), and ischemia-driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Stent thrombosis (ST) | 5-years
  Thrombosis of the stent after PCI
Intrastent-restenosis (ISR) | 5-years
  Intrastent restenosis with >50% of the stent diameter
Target Vessel MI (TVMI) | 5-years
  Target vessel myocardial infarction at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Rivoli Hospital, Rivoli, Turin, Italy

IPD SHARING:
Plan to Share IPD: No